CLINICAL TRIAL: NCT00853814
Title: Increasing Youth Physical Activity: Neighborhood Environment Influences
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: James N. Roemmich, Associate Professor of Pediatrics, University at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD055270 (NIH); 5R01HD055270-02 (NIH); 5R01HD055270-03 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2009-03-02 (Estimated); Status verified 2009-02

CONDITIONS: Obesity; Overweight
Keywords: adolescence; obesity; physical activity; built environment; neighborhood environment; children; youth; increasing physical activity; changing dietary intake; reducing zBMI
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Reduced access to sedentary behaviors, High park access (Experimental)
  Interventions: Behavioral: Access to sedentary behaviors
- Usual access to sedentary behaviors, High park access (Experimental)
  Interventions: Behavioral: Access to sedentary behaviors
- Reduced access to sedentary behaviors, Low park access (Experimental)
  Interventions: Behavioral: Access to sedentary behaviors
- Usual access to sedentary behaviors, Low park access (Experimental)
  Interventions: Behavioral: Access to sedentary behaviors

INTERVENTIONS:
Behavioral: Access to sedentary behaviors — Access to sedentary behaviors: Reduced access - reduce access to sedentary behaviors by 50% using TV Allowance technology. Usual access - monitoring only, no change in access to sedentary behaviors. Access to neighborhood parks: High access - large amount of park land very near to the child's home. Low access - little to no park land near the child's home.

SUMMARY:
Increased access to highly reinforcing sedentary behaviors in the home such as TV and computers are associated with overweight in youth. Reducing these behaviors reduces overweight and prevents increases in overweight in youth who are at risk, likely by increasing physical activity and/or reducing energy intake. Reducing access to highly reinforcing sedentary activities frees-up time and youth must choose to reallocate their time between engaging in other, less reinforcing sedentary activities or physical activity. Neighborhood environments that provide easy access to reinforcing physical activities such as those at parks may result in greater increases in physical activity when access to highly reinforcing home sedentary behaviors is reduced. The investigators have found in 3 data sets of youth ranging in age from 4 to 16 years that the proportion of park and recreation area to residential area within ½ mile of the child's home parcel (park and recreation index) independently predicted the physical activity of youth. The investigators also found that increases in physical activity when access to sedentary behaviors were reduced for 3 weeks was related to park area within ½ mile of the child's home. The aim of this study is to decrease access to home sedentary behaviors for 4 months and determine if changes in physical activity habits are related to access to parks and recreation areas in the neighborhood environment. The investigators propose to study 128 sedentary overweight male and female 12-14 year-old youth recruited from parcels within Erie County, New York that have a high or low park and recreation index. Groups will be matched on racial/ethnic distribution and socioeconomic status. Subjects living at low and high park access parcels will then be equally randomized to groups that reduce targeted sedentary behavior (TV, computer use) time by 50% using TV Allowance devices placed on each TV/monitor in the home or a control group that has the same experimental experiences including TV Allowance devices placed on each TV/monitor, but programmed to not limit access to targeted sedentary behavior. Subjects will wear both accelerometers and wrist-watch-type global positioning systems to determine changes in the duration and intensity of physical activity in various parcel types, including parks. The investigators hypothesize differential responses in physical activity and the utilization of parks for physical activity. The group of youth that live at parcels with high access to parks and that incur a 50% reduction in sedentary behavior will have greater increases in physical activity, number of visits to parks and will accrue greater physical activity at parks than youth in the other 3 treatment groups. The investigators hypothesize that the alterations in physical activity will be mediated by parent modeling of physical activity and individual differences in the motivation to be physically active. The investigators hypothesize that there will be a main effect of reduction in access to sedentary behaviors on energy and fat intake and percent overweight.

ELIGIBILITY:
Inclusion Criteria:

* Parent and child must wear an accelerometer and record their sedentary behaviors
* Youth must engage in at least 24 h/week of time in sedentary behaviors
* Youth should have no dietary or activity restrictions
* Youth and parents should have no psychopathology that would limit participation
* No contraindications to physical activity in either the parent or adolescent

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 10 weeks

SECONDARY OUTCOMES:
Physical activity in parks | 10 weeks
Dietary intake | 10 weeks
BMI percentile | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James N Roemmich, Ph.D., Principal Investigator — University at Buffalo; Samina Raja, Ph.D., Principal Investigator — University at Buffalo; Leonard H Epstein, Ph.D., Principal Investigator — University at Buffalo; Li Yin, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States